CLINICAL TRIAL: NCT02866292
Title: Is There Relationship Between the Pelvic Floor Muscles Strength and Sexual Function in Primigravid and Non-pregnant Nulliparous?
Brief Title: The Pelvic Floor Muscles Strength and Sexual Function in Primigravid and Non-pregnant Nulliparous
Status: Completed | Type: Observational
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Marília Duarte dos Santos, Principal Investigator, Federal University of Uberlandia
Other Study IDs: CEP UFU 145.623/2012
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Sexual Behavior
Keywords: Pelvic Floor; Pregnancy; Physical Therapy Specialty
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- non-pregnant nulliparous: Nulliparous without previous gestation. Pelvic floor muscle evaluation by means of vaginal palpation and vaginal squeeze pressure (perineometer), and evaluation of the sexual function by the Female Sexual Function Index (FSFI) questionnaire.
  Interventions: Other: Pelvic floor muscle and sexual function evaluation
- primigravid: Pregnant women on her first pregnancy and gestational age above 14 weeks. Pelvic floor muscle evaluation by means of vaginal palpation and vaginal squeeze pressure (perineometer), and evaluation of the sexual function by the Female Sexual Function Index (FSFI) questionnaire.
  Interventions: Other: Pelvic floor muscle and sexual function evaluation

INTERVENTIONS:
Other: Pelvic floor muscle and sexual function evaluation — PFM evaluation was performed by vaginal palpation and vaginal squeeze pressure. During vaginal palpation the physiotherapist introduced the index and middle fingers about 4cm inside the vagina, and requested to hold the maximum contraction of the PFM. Muscle function was classified by the Oxford Scale Modified.
  The vaginal squeeze pressure was measured through Perineometer.To obtain the measurements, the subjects remained positioning and vaginal sensor was introduced into the vaginal cavity. The women were oriented and motivated verbally to perform three voluntary maximal contractions sustained for five seconds and one minute interval between them.
  Sexual function was evaluated by the Female Sexual Function Index (FSFI) questionnaire. The questionnaire consists of 19 multiple-choice questions, which involves six sexual response domains: desire, arousal, lubrication, orgasm, satisfaction and pain.

SUMMARY:
This study has two aims: a) to evaluate the pelvic floor muscles strength in primigravid and non-pregnant nulliparous women and to correlate with their sexual function and b) to compare PFM strength and sexual function between women in the second and third pregnancy trimesters.

DETAILED DESCRIPTION:
This is an observational cross-sectional study. The sample consisted of 161 women divided into two groups: the first of pregnant women, formed by 81 primigravidae participants in the Prenatal Program of the public health system in Uberlandia city (Brazil). The second consists of 80 non-pregnant nulliparous. All participants signed an informed consent and the study was approved by the Ethics Committee of the Federal University of Uberlandia (nº 145.623/2012).

To estimate the average strength of vaginal palpation and vaginal squeeze pressure in primigravid, the investigators used the following equation to scale the sample: Zα/2 refers to the probability (α/2) standard one-tailed normal distribution; σ2 is the variance associated with vaginal palpation and vaginal squeeze pressure; ε is the sampling error. Based on a similar study, which evaluated similar population, it was assumed: α=0.05, σ=1.34 and ε=0.32 for vaginal palpation; and it was assumed: α=0.05, σ=12.60 and ε=3.00 for vaginal squeeze pressure. Therefore, the sample size would be 67 and 68 women, respectively.

The PFM assessment

PFM evaluation was performed by vaginal palpation and vaginal squeeze pressure. These methods are widely used in research involving the female pelvic floor and many studies have shown its reproducibility and validity.

The same examiner conducted all evaluations and before the start of the study, the reproducibility was tested. Ten women were evaluated twice, with an interval of one week to determine the intraclass correlation coefficient (ICC) of all variables.

The participants were asked about the health history. After checking that they were eligible to participate in the survey, participants were invited to empty the bladder and to remain in the supine position with hips and knees flexed and feet propped. Assessments began after explaining how to perform the contraction of PFM and the volunteer was advised to stay relaxed and breathing normally. The vaginal palpation was always the first exam to check the PFM contraction ability and then was held vaginal squeeze pressure exam.

During vaginal palpation the examiner quantified strength. The physiotherapist introduced the index and middle fingers about 4cm inside the vagina, and requested to hold the maximum contraction of the PFM, according to the instruction of a movement "inward and up" with the greatest possible strength. Muscle function was classified by the Oxford Scale Modified, with varies from zero (absence of muscle contraction) to five (strong contraction with finger sucking of the evaluator). To be considered valid, the movement of cranial elevation was observed by the examiner, as well as the absence of visible contractions of the adductor muscles of the hip, gluteus or abdominals.

The vaginal squeeze pressure was measured through perineometer equipped with a vaginal probe that has been covered with a non-lubricated condom and then the probe was lubricated with hypoallergenic gel. The probe sensor was connected to a microprocessor hand with a latex tube, which allows the measurement of nip pressure in centimeters of water. To obtain the measurements, the subjects remained positioning and vaginal sensor was introduced approximately 4cm into the vaginal cavity. The women were oriented and motivated verbally to perform three voluntary maximal contractions sustained for five seconds and one minute interval between them. For statistical analysis, the investigators used the mean of three peak pressures provided by the equipment.

Sexual function assessment

Sexual function was evaluated by the Female Sexual Function Index (FSFI) questionnaire, with a validated Portuguese version, which has an easy to understand language and subsequently was applied exclusively in Brazilian pregnant women. The questionnaire consists of 19 multiple-choice questions, which involves six sexual response domains: desire, arousal, lubrication, orgasm, satisfaction and pain. The score for each question is individual, varying from 0 to 6 points. The investigators performed a mathematical calculation, which allowed the acquisition of a ﬁnal index, the total score of the FSFI. The total score of FSFI ranges between 2 and 36 points. The lower the score, the worse is the sexual function is. The assessment is for the period of the last four weeks.

At the time of the interview, the pregnant women were instructed regarding the completion and they had their enough time to fill it out in a self-administered way in a reserved place.

Statistical analysis

Statistical analysis was performed using Statistical Package for Social Sciences software (SPSSV21, Chicago, IL). Data normality was tested by the Kolmogorov-Smirnov test. To perform the variables comparison, the Mann-Whitney test was performed. To verify the correlation between the variables, the Spearman correlation test was used. Values of p<0.05 were considered significant. The intensity of the relationship of the correlation coefficient values were interpreted according to the following guidelines: 0 = zero; 0.10-0.39 = weak; 0.40-0.69 = moderate; 0.70-0.99 = strong, 1 = perfect, regardless of whether positive or negative.

ELIGIBILITY:
Inclusion Criteria:

* Be non-pregnant nulliparous or primigravid women with pregnant only one fetus alive and without abnormalities that could increase uterine volume
* Present ability to contract the pelvic floor muscles
* Report at least one sexual relationship in the four weeks prior to data collection

Exclusion Criteria:

* Were previous urogynecological surgery history
* Non-pregnant nulliparous who did not have sexual intercourse with vaginal penetration
* Presence of cognitive impairment or neurological condition that could affect muscle activation
* Present urinary tract infection at the time of data collection.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The sample consisted of 154 women divided into two groups: the first of pregnant women, formed by 76 primigravidae participants in the Prenatal Program of the public health system in Uberlandia city (Brazil). The second consists of 78 non-pregnant nulliparous.
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2014-11; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
muscle strength with Oxford scale | through study completion, an average of 1 year
score of Female Sexual Function Index questionnaire | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Marília Duarte dos Santos, Uberlândia, Minas Gerais, Brazil

REFERENCES:
- [Background] Pereira VS, Hirakawa HS, Oliveira AB, Driusso P. Relationship among vaginal palpation, vaginal squeeze pressure, electromyographic and ultrasonographic variables of female pelvic floor muscles. Braz J Phys Ther. 2014 Sep-Oct;18(5):428-34. doi: 10.1590/bjpt-rbf.2014.0038. Epub 2014 Oct 10. PMID 25372005
- [Result] Bo K, Finckenhagen HB. Vaginal palpation of pelvic floor muscle strength: inter-test reproducibility and comparison between palpation and vaginal squeeze pressure. Acta Obstet Gynecol Scand. 2001 Oct;80(10):883-7. doi: 10.1034/j.1600-0412.2001.801003.x. PMID 11580731
- [Result] Arab AM, Behbahani RB, Lorestani L, Azari A. Correlation of digital palpation and transabdominal ultrasound for assessment of pelvic floor muscle contraction. J Man Manip Ther. 2009;17(3):e75-9. doi: 10.1179/jmt.2009.17.3.75E. PMID 20046616